CLINICAL TRIAL: NCT07069400
Title: An International Observational Study of Adults With Acute Infection
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STRIVE 002
Record Dates: First submitted 2025-05-12; First posted 2025-07-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, blood, whole blood, nasal swab, urine, sputum, tracheal aspirate, stool or rectal swab, and skin lesion sampling.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: The study population includes adult patients admitted to a hospital with a suspected or confirmed acute infection.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
Prospective, longitudinal studies of people with acute infections are essential to understand risk factors, clinical manifestations, pathobiology, and management strategies. Observational studies can provide data necessary to select interventions and strategies for testing in clinical trials and to develop key design features of trials. Observational studies can be particularly important for establishing an early knowledge base after emergence of a new pathogen, as illustrated by the recent emergence of influenza A (H1N1), SARS-CoV-2, and Mpox. This observational study protocol describes collection of data and biospecimens from sites across the world for characterizing acute infections in hospitalized patients. The protocol is designed to study respiratory infections, infections outside the respiratory tract, established infectious diseases, and emerging infectious diseases. Data generated in this study will be used to efficiently characterize acute infectious diseases and plan future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Admitted to hospital (or in an emergency department with anticipated hospital admission) for the management of a suspected or confirmed acute infectious disease.
* Onset of symptoms of an infectious disease within the past 30 days.
* Informed consent for study participation by the participant or a surrogate decision maker if the participant lacks capacity for consent.

Exclusion Criteria:

* Current imprisonment (this does not include quarantine for an infectious disease).
* Patient undergoing comfort care measures only such that treatment focuses on end- of-life symptom management over prolongation of life.
* Expected inability or unwillingness to participate in study procedures.
* In the opinion of the investigator, participation in the study is not in the best interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled at study sites globally. Study personnel at the enrolling site will confirm eligibility and obtain consent prior to beginning study procedures. Signing of the informed consent document signifies study entry and Study Day 0. The study population includes adult patients admitted to a hospital with a suspected or confirmed acute infection. All participants will meet the eligibility criteria below. Specific studies executed with this master protocol may narrow the eligibility criteria to a more specific population (that is, a subset of patients who meet the eligibility criteria in this overarching protocol).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2027-06-08 (Estimated); Study Completion 2027-06-08 (Estimated)

PRIMARY OUTCOMES:
Day 28 Mortality | Day 28
  All-cause mortality
Days to recovery scale (DRS) | Day 28
  The Days to Recovery Scale (DRS) is an ordinal ranked outcome that includes the concepts of mortality and time to recovery, with recovery defined as being discharged from the hospital and reaching home for the duration of the follow- up. At the end of the follow-up period, each patient is classified into one of the DRS categories based on vital status, hospitalization status, and duration it took to reach recovery.
Time to Sustained Recovery | Day 28
  Time to sustained recovery is defined as being discharged from the index hospitalization, followed by being alive and home for 14 days.
Ordinal outcome for clinical improvement - Day 7 | Day 7
  For respiratory infections, the WHO Ordinal Scale for Clinical Improvement may be assessed.
Organ support free days | Day 28
  the number of days between enrollment and hospital discharge or day 28 that the participant did not receive support for some organ (lungs, kidneys, etc.)
The Sequential Organ Failure Assessment (SOFA) score - Day 28 | Day 28
  The SOFA score is one of the most widely used scoring systems in critically ill patients and has also been validated in hospitalized patients with suspected infection outside the ICU. This score assesses organ dysfunction across 6 organ systems. To facilitate use of the SOFA score across a broad range of sites, including those in low- and-middle income countries (LMICs), SpO2 may be substituted for PaO2, and the presence of scleral icterus or jaundice may be substituted for serum bilirubin level . Only clinically available data will be used to calculate SOFA scores. Laboratory tests will not be completed by the study to calculate SOFA scores.

CONTACTS AND LOCATIONS:
Overall Officials: Cavan Reilly, PhD, Principal Investigator — University of Minnesota
Locations (28):
- United States (10):
  - Stanford University Hospital & Clinics (Site 203-003), Palo Alto, California
  - UCSF Medical Center (Site 203-001), San Francisco, California
  - University of Kansas Medical Center (Site 080-044), Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Mount Sinai Medical Center (Site 301-012), New York, New York
  - Wake Forest Baptist Health (210-001), Winston-Salem, North Carolina
  - Cleveland Clinic Foundation (Site 207-001), Cleveland, Ohio
  - Vanderbilt University Medical Center (Site 212-001), Nashville, Tennessee
  - UT Southwestern Medical Center (084-001), Dallas, Texas
  - Intermountain Medical Center (Site 211-001), Murray, Utah
- Hospital General de Agudos JM Ramos Mejia (Site 611-001), Buenos Aires, Argentina
- Australia (2):
  - St. Vincent's Hospital (612-002), Sydney, New South Wales
  - Royal Brisbane and Women's Hospital (Site 612-055), Brisbane, Queensland
- CERMIPA (Site 403-001), Abidjan, Côte d’Ivoire
- Rigshospitalet, CHIP (625-006), Copenhagen, Denmark
- Greece (2):
  - Evangelismos General Hospital (Site 635-020), Athens, Attica
  - 3rd Dept of Medicine, Medical School (Site 635-022), Athens, Attica
- Japan (2):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Japan Institute for Health Security, Tokyo
- Tan Tock Seng Hospital, Singapore, Singapore
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul St. Mary's Hospital, Seoul
- Hospital Universitari Germans Trias i Pujol (Site 626-003), Badalona, Barcelona, Spain
- Chulalongkorn University and The HIV-NAT (Site 613-001), Bangkok, Thailand
- Uganda (2):
  - MRC/UVRI & LSHTM Uganda Research Unit (Site 634-601), Entebbe
  - Lira Regional Referral Hospital (Site 634-605), Lira
- Central City Clinical Hospital of Ivano-Frankivsk City Council (627-302), Ivano-Frankivsk, Ukraine
- Royal Free Hospital (Site 634-006), London, United Kingdom